CLINICAL TRIAL: NCT01852422
Title: Location and Anatomic Characterization of the Sacrospinous Ligaments in Women With Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Pop Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: POP protocol 01
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pelvic prolapse

SUMMARY:
Pelvic organ prolapse is a common disorder that results in significant patient morbidity. Approximately 1 in 9 women undergo surgery for the correction of pelvic organ prolapse (POP) and associated bladder and bowel dysfunction. Despite its common occurrence, the cause of POP remains largely unknown. Prolapse is thought to be caused by direct injury to the levator ani (LA) muscle, denervation of the pelvic floor musculature, or fascial damage incurred during childbirth trauma. The sacrospinous ligaments are commonly employed surgical structures employed to repair vaginal prolapse. Despite the frequent use of these structures in prolapse surgery, there is a paucity of information regarding the identification of these structures outside of surgical dissection. Furthermore, there is no published data describing the relative distances between the apex of the vagina and these ligaments in women with prolapse. Recent developments in imaging have enabled the identification of the distal subdivisions of the levator ani, classifying as: pubovaginalis, puboanalis, and the puboperinealis as the subdivisions of the pubovisceralis. The visualization of these structures is possible using a 3D ultrasound technique (BK medical, Wilmington, MA), that has been validated in cadavers and in live humans, with excellent interrater reliability. The investigators propose to use this technology to explore the anatomy of the sacrospinous ligaments.

ELIGIBILITY:
Inclusion Criteria:

* age 21-80 years old
* Stage III or higher pelvic prolapse

Exclusion Criteria:

-Prior pelvic surgery

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pelvic organ prolapse 21-80 years old
Sampling Method: Non-Probability Sample
Dates: Start 2013-06; Primary Completion 2013-08-03 (Actual); Study Completion 2023-10-30

PRIMARY OUTCOMES:
Unequivocal identification of the sacrospinous ligaments, in real time, by ultrasound imaging | Real time during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee MC, Nahariya, Israel